CLINICAL TRIAL: NCT04142775
Title: Predictors of Intracranial Hemorrhage in Critically Ill Patients With Acute Lung Failure (ARDS) on Extracorporeal Membrane Oxygenation (ECMO)
Brief Title: Predictors of Intracranial Hemorrhage in ARDS Patients on ECMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Mario Menk, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: ChariteMM
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: ARDS, Human; Extracorporeal Membrane Oxygenation Complication
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- intracranial hemorrhage (ICH): ARDS patients treated with ECMO developing ICH
  Interventions: Other: complication versus no complication
- no intracranial hemorrhage: ARDS patients treated with ECMO not developing ICH

INTERVENTIONS:
Other: complication versus no complication — development of ICH
  Groups: intracranial hemorrhage (ICH)

SUMMARY:
Intracranial hemorrhage is is a rare, but critical incident in patients with acute lung failure undergoing ECMO therapy. Predictors of intracranial hemorrhage are yet to be defined to identify patients at (high) risk. This retrospective analysis investigates the predictive value and validity of parameters and specific risk factors of critically ill ARDS patients treated with ECMO.

ELIGIBILITY:
Inclusion Criteria:

* ARDS following Berlin definition (mild, moderate, severe)
* ECMO therapy (veno-venous cannulation)

Exclusion Criteria:

* ECMO, other than VV
* ICH at initiation of ECMO
* no cerebral CT scan at any time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill patients on the ICU with acute lung failure (ARDS) in a German regional ARDS referral center
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
mortality | up to 28 days
  mortality after ICH/no ICH in ARDS patients with ECMO

SECONDARY OUTCOMES:
ICU stay | up to 28 days
  days on ICU
ventilator/ECMO-free days | up to 28 days
  Ventilator/ECMO-free days

CONTACTS AND LOCATIONS:
Locations (1):
- Charite university medicine Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No